CLINICAL TRIAL: NCT06235411
Title: Psilocybin in Alcohol Use Disorder With Comorbid Depression
Acronym: PAD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IRESP/2022/AL-01
Record Dates: First submitted 2024-01-08; First posted 2024-01-31 (Actual); Last update posted 2025-03-19 (Actual); Status verified 2025-03

CONDITIONS: Alcohol-Related Disorders; Depressive Disorder; Addiction
Keywords: Psilocybin; Psychedelic assisted therapy
MeSH Terms: conditions — Alcohol-Related Disorders; Depressive Disorder; Behavior, Addictive | interventions — Blood Specimen Collection

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental group (Experimental)
  Interventions: Drug: Psilocybin therapy; Other: Electroencephalogram; Other: Blood samples for the analysis of immune and inflammatory profiles; Other: stool samples; Other: MRI functional and cerebral
- Control group (Placebo Comparator)
  Interventions: Drug: Inactive Psilocybin therapy; Other: Electroencephalogram; Other: Blood samples for the analysis of immune and inflammatory profiles; Other: stool samples; Other: MRI functional and cerebral

INTERVENTIONS:
Drug: Psilocybin therapy — Two administrations of psilocybin given 3 weeks apart. The treatment day will begin around 9 a.m. with a brief interview. Patients will be invited to relax and music will be played through speakers and headphones.
  One 25 mg capsule of Psilocybin will be given approximately 30 minutes to 1.5 hours later.
  The patient is accompanied throughout the session (minimum 6 hours depending on the effects felt). The patient will benefit from a preparation session the day before dosing, and an integration session the day after. Intensive relapse prevention program will be dispensed between the 2 dosing sessions (treatment as usual).
  Arms: Experimental group
Drug: Inactive Psilocybin therapy — Two administrations of psilocybin given 3 weeks apart. The treatment day will begin around 9 a.m. with a brief interview. Patients will be invited to relax and music will be played through speakers and headphones.
  One 1 mg capsule of Psilocybin will be given approximately 30 minutes to 1.5 hours later.
  The patient is accompanied throughout the session (minimum 6 hours depending on the effects felt). The patient will benefit from a preparation session the day before dosing, and an integration session the day after. Intensive relapse prevention program will be dispensed between the 2 dosing sessions (treatment as usual).
  Arms: Control group
Other: Electroencephalogram — * Rest EEG prior to first treatment administration
  * EEG during first treatment administration
  * Rest EEG during integration session after second treatment administration
Other: Blood samples for the analysis of immune and inflammatory profiles — Three 7ml EDTA tubes will be taken in the morning on an empty stomach at day 0 and at 3 weeks.
Other: stool samples — Stool sampling at day 0 and 3 weeks Analysis of intestinal microbiota is carried out on a stool sample, which is stored at -20°C for a maximum of 24 hours. The sample is then transferred cold to the CRB of the Nîmes University Hospital, where it is stored at -80°C until the microbiology laboratory can perform a group analysis.
Other: MRI functional and cerebral — MRI functional and cerebral at day 0 and 3 weeks

SUMMARY:
Up to 40% of people with alcohol use disorder (AUD) experience depression. Depression is a risk factor for early relapse of AUD after withdrawal in a controlled environment. Promising data suggest the effectiveness of psilocybin, a psychedelic-type treatment, in depression and AUD. Following the acute effects of the psychedelic experience, which lasts approximately 6 hours, psilocybin action appears to be beneficial for preventing alcohol relapse in recently weaned people suffering from comorbid depression. Whilst the public perception of psilocybin therapy is poorly documented in France, the rapid changes in the legal status of psilocybin elsewhere, the positive media coverage of recent trials in depression, and the recent designation as an "innovative therapy" by the FDA could lead to the refusal of randomization of eligible participants. It is therefore essential to evaluate the feasibility and acceptability of psilocybin treatment and blinded randomized design in our clinical population of hospitalized patients with AUD and depressive symptoms. Recent data suggest that the effect size of psilocybin is much higher than other currently available treatments. However, this paradigm shift must be confirmed in our cohort of people with AUD and depressive symptoms, and in the context of treatment in addition to usual care, by an estimation of the expected effect size based on real data. This will allow the sample size to be accurately calculated for a large-scale randomized clinical trial. Finally, the potential mechanisms of action of psilocybin to prevent relapse in AUD with comorbid depression after withdrawal need to be documented. The objective of this pilot study is to evaluate the feasibility, acceptability, neural mechanisms and preliminary results of the effectiveness of psilocybin in the treatment of AUD and depressive symptoms after withdrawal, in addition to usual treatment. The study authors hypothesize that two oral administrations of 25 mg psilocybin at three-week intervals versus a control condition (1 mg psilocybin), in addition to the usual treatment, will be acceptable and feasible in recently withdrawn individuals suffering from AUD and depressive symptoms, between 14 and 60 days after their last alcohol consumption

ELIGIBILITY:
Inclusion Criteria:

* Patient with a confirmed DSM-5 diagnosis of severe alcohol use disorder.
* BDI II (Beck Depression Inventory) score ≥ 14.
* Last alcohol consumption must have occurred between 60 and 14 days prior to study inclusion. The patient must have had at least one heavy drinking day during the last period of alcohol consumption.

NB: The last period of alcohol consumption prior to inclusion is defined as the last 4 weeks counted from the last drink.

* Patient with free and informed consent.
* The patient must be a member or beneficiary of a health insurance plan

Exclusion Criteria:

* The subject is participating in an interventional study involving a drug or in a clinical trial according to the REC.
* The subject is in a period of exclusion determined by a previous study
* The subject unable to express consent
* It is impossible to give the subject informed information
* The patient is under safeguard of justice or state guardianship
* Schizophrenic disorder, or any history of psychotic disorder according to the clinician's judgment.
* Past or current manic or hypomanic episode.
* Need for antipsychotic treatment that may interfere with psilocybin.
* Need for treatment with monoamine oxidase inhibitors (MAOIs) which may interfere with psilocybin.
* Current scripted suicidal ideation (according to clinician judgment) corresponding to a "high risk" score on the Columbia-Suicide Severity Rating Scale (C-SSRS).
* First-degree family member diagnosed with psychotic disorder or bipolar disorder type 1.
* High risk of negative emotional or behavioral response based on the investigator's clinical judgment (e.g., signs of serious personality disorders, antisocial behavior, severe current stressors, lack of meaningful social support)
* Patient with dementia or severe cognitive impairment (as judged by the clinician).
* CIWA-R score ≥ 8.
* Medical conditions that would prevent safe participation in the trial; for example: seizure disorders, significant impairment of liver function, coronary heart disease, history of arrhythmia, heart failure, uncontrolled hypertension (greater than 165/95 mmHg at screening), history of stroke, severe asthma, hyperthyroidism, narrow-angle glaucoma, stenotic peptic ulcer, pyloroduodenal obstruction, symptomatic enlarged prostate or bladder neck obstruction), Uncontrolled type I or type II diabetes or history of ketoacidosis, hyperglycemic coma or severe hypoglycemia with loss of conscience
* History of hallucinogen use disorder, any use in the past year or >25 lifetime uses.
* Dependence on cocaine, psychostimulants, opioids or cannabis (last 12 months).
* Current non-medical use of cocaine, psychostimulants or opioids (past 30 days).
* Serious ECG abnormalities (e.g., signs of ischemia, myocardial infarction, QTc prolongation (QTc > 0.45 seconds for men, QTc > 0.47 seconds for women).
* Hypersensitivity to the active ingredient or excipients
* No access to email.
* Insufficient understanding of French to complete the questionnaires.
* Patient for whom it is impossible to provide informed information.
* Pregnant or breastfeeding patient.
* Patient planning a pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2024-02-05 (Actual); Primary Completion 2024-11-19 (Actual); Study Completion 2025-01-09 (Actual)

PRIMARY OUTCOMES:
Feasibility of the intervention between groups | After 2nd experimental session (Week 4)
  Number of patients who completed both sessions

SECONDARY OUTCOMES:
Feasibility of recruitment between groups | 18 Months
  Number of patients screened per month/number of patients included per month.
Feasibility of retainment between groups | 18 Months
  Average time (days) between screening and inclusion.
Feasibility of the trial between groups | 18 Months
  Rate (%) of eligible patients who are included in the study.
Feasibility of randomization between groups | 18 Months
  Rate (%) of patients included who had at least one treatment administration session
Feasibility of inclusion between groups | 18 Months
  Rate (%) of assessment sessions that were completed.
Feasibility of therapeutic intervention between groups | 18 Months
  Duration of assessment sessions (minutes).
Study acceptability between groups | 18 Months
  Number of patients leaving the study prematurely for any reason.
Patient-reported reasons for abandoning the study between groups | 18 Months
  Qualitative description of reasons cited by patients
Decrease in alcohol consumption between groups | Day 0
  Decrease in the percentage of days of heavy drinking days during previous 4 weeks versus baseline
Decrease in alcohol consumption between groups | Week 6 (or discharge if it takes place later)
  Decrease in the percentage of days of heavy drinking days during previous 4 weeks versus baseline
Decrease in alcohol consumption between groups | Week 12
  Decrease in the percentage of days of heavy drinking days during previous 4 weeks versus baseline
Total alcohol consumption between groups | Day 0
  Total alcohol consumption during previous 4 weeks
Total alcohol consumption between groups | Week 6 (or discharge if it takes place later)
  Total alcohol consumption during previous 4 weeks
Total alcohol consumption between groups | Week 12
  Total alcohol consumption during previous 4 weeks
Time before first drink | Day 0
  Days
Time before first drink | Week 6 (or discharge if it takes place later)
  Days
Time before first drink | Week 12
  Days
Time to first day of heavy drinking | Day 0
  Days
Time to first day of heavy drinking | Week 6 (or discharge if it takes place later)
  Days
Time to first day of heavy drinking | Week 12
  Days
Craving between groups | Day 0
  Craving Experience Questionnaire (CEQ) score; the CEQ evaluates intensity and frequency of craving from 11 intensity items in blocks a-c. Each item is rated between 0 ("Not at all") and 10 ("Extremely") for a total score between 0 and 110. The higher the score, the more intense the craving. A frequency of craving score is calculated by adding the values obtained from 11 items in blocks d-f. Each item is rated between 0 ("Never") and 10 ("Constantly") for a total craving frequency score between 0 and 110.
Craving between groups | Week 12
  Craving Experience Questionnaire (CEQ) score; the CEQ evaluates intensity and frequency of craving from 11 intensity items in blocks a-c. Each item is rated between 0 ("Not at all") and 10 ("Extremely") for a total score between 0 and 110. The higher the score, the more intense the craving. A frequency of craving score is calculated by adding the values obtained from 11 items in blocks d-f. Each item is rated between 0 ("Never") and 10 ("Constantly") for a total craving frequency score between 0 and 110.
Quality of life between groups | Day 0
  Alcohol quality of life scale (AQoLS); the 34-item questionnaire measures the negative impact of the relationship with alcohol on quality of life through 7 dimensions: social relationships, activities, living conditions, etc. self-care, negative emotions, sleep and loss of control on a scale of 0 (not at all) to 3 (very much), for a total score of 102. There is no threshold value.
Quality of life between groups | Week 12
  Alcohol quality of life scale (AQoLS); the 34-item questionnaire measures the negative impact of the relationship with alcohol on quality of life through 7 dimensions: social relationships, activities, living conditions, etc. self-care, negative emotions, sleep and loss of control on a scale of 0 (not at all) to 3 (very much), for a total score of 102. There is no threshold value.
Depression between groups | Day 0
  Beck Depression Inventory (BDI II); a 21-item scale. Each item consists of 4 sentences corresponding to 4 degrees of increasing intensity of a symptom, rated from 0 to 3. Only the highest rating chosen for a given series is retained. The total score ranges from 0 to 39; with a higher score indicating greater intensity of depression.
Depression between groups | Week 12
  Beck Depression Inventory (BDI II); a 21-item scale. Each item consists of 4 sentences corresponding to 4 degrees of increasing intensity of a symptom, rated from 0 to 3. Only the highest rating chosen for a given series is retained. The total score ranges from 0 to 39; with a higher score indicating greater intensity of depression.
Anxiety between groups | Day 0
  Beck Anxiety Inventory (BAI); a 21-question score of common symptoms of anxiety, such as numbness and tingling, and sweating. Responses are rated on a scale of 0 (not at all) to 3 (severely). Higher total scores indicate more severe anxiety symptoms. Thresholds are: 0-7: Minimal; 8-15: Light; 16-25: Moderate; 26-63: Severe.
Anxiety between groups | Week 12
  Beck Anxiety Inventory (BAI); a 21-question score of common symptoms of anxiety, such as numbness and tingling, and sweating. Responses are rated on a scale of 0 (not at all) to 3 (severely). Higher total scores indicate more severe anxiety symptoms. Thresholds are: 0-7: Minimal; 8-15: Light; 16-25: Moderate; 26-63: Severe.
Emotion regulation difficulties between groups | Day 0
  Difficulties in Emotion Regulation Scale (DERS); a 36-item questionnaire assessing multiple aspects of emotion dysregulation. The measure gives a total score and six subscores:1. Non-acceptance of emotional responses (NON-ACCEPTANCE); 2. Difficulties in adopting goal-oriented behavior (GOALS); 3. Difficulty controlling impulses (IMPULSE); 4. Lack of emotional awareness (AWARENESS); 5. Limited access to emotion regulation strategies (STRATEGIES); 6. Lack of emotional clarity (CLARITY), with a final score 0-100.
Emotion regulation difficulties between groups | Week 12
  Difficulties in Emotion Regulation Scale (DERS); a 36-item questionnaire assessing multiple aspects of emotion dysregulation. The measure gives a total score and six subscores:1. Non-acceptance of emotional responses (NON-ACCEPTANCE); 2. Difficulties in adopting goal-oriented behavior (GOALS); 3. Difficulty controlling impulses (IMPULSE); 4. Lack of emotional awareness (AWARENESS); 5. Limited access to emotion regulation strategies (STRATEGIES); 6. Lack of emotional clarity (CLARITY), with a final score 0-100.
Rejection sensitivity between groups | Day 0
  Adult Rejection Sensitivity Questionnaire (A-RSQ); rejection sensitivity score calculated for 9 situations by multiplying the level of rejection concern by the level of rejection expectation. The total rejection sensitivity score is the average of the rejection sensitivity scores for the 9 situations.
Rejection sensitivity between groups | Week 12
  Adult Rejection Sensitivity Questionnaire (A-RSQ); rejection sensitivity score calculated for 9 situations by multiplying the level of rejection concern by the level of rejection expectation. The total rejection sensitivity score is the average of the rejection sensitivity scores for the 9 situations.
Meaning in life between groups | Day 0
  Meaning in Life Questionnaire (MLQ); a 10-item score assessing two dimensions of meaning in life rated on a seven-point scale ranging from "absolutely true" to "absolutely false." The "Presence of Meaning" subscale measures the extent to which respondents believe their lives have meaning. The "Search for Meaning" subscale measures respondents' engagement and motivation in their efforts to find meaning or deepen their understanding of the meaning of their lives, with a final score of 5-35
Meaning in life between groups | Week 3
  Meaning in Life Questionnaire (MLQ); a 10-item score assessing two dimensions of meaning in life rated on a seven-point scale ranging from "absolutely true" to "absolutely false." The "Presence of Meaning" subscale measures the extent to which respondents believe their lives have meaning. The "Search for Meaning" subscale measures respondents' engagement and motivation in their efforts to find meaning or deepen their understanding of the meaning of their lives, with a final score of 5-35
Meaning in life between groups | Week 6
  Meaning in Life Questionnaire (MLQ); a 10-item score assessing two dimensions of meaning in life rated on a seven-point scale ranging from "absolutely true" to "absolutely false." The "Presence of Meaning" subscale measures the extent to which respondents believe their lives have meaning. The "Search for Meaning" subscale measures respondents' engagement and motivation in their efforts to find meaning or deepen their understanding of the meaning of their lives, with a final score of 5-35
Meaning in life between groups | Week 12
  Meaning in Life Questionnaire (MLQ); a 10-item score assessing two dimensions of meaning in life rated on a seven-point scale ranging from "absolutely true" to "absolutely false." The "Presence of Meaning" subscale measures the extent to which respondents believe their lives have meaning. The "Search for Meaning" subscale measures respondents' engagement and motivation in their efforts to find meaning or deepen their understanding of the meaning of their lives, with a final score of 5-35
Cognitive functioning between groups | Day 0
  Conflict indices and task focus of the Visual Perspective Task (VPT); participants evaluate either the number of red dots that in a scene from their own point of view (self-perspective condition), or the number of dots that another no one present in the scene can see (self-perspective condition).
Cognitive functioning between groups | Second psilocybin session (Week 4)
  Conflict indices and task focus of the Visual Perspective Task (VPT); participants evaluate either the number of red dots that in a scene from their own point of view (self-perspective condition), or the number of dots that another no one present in the scene can see (self-perspective condition).
Role of cognitive function at baseline on change in the percentage of heavy drinking days in preceding 4 weeks | Day 0
  Montreal Cognitive Assessment (MoCA); measuring attention, concentration, executive functions, memory, language, visuoconstructive abilities, abstraction abilities, calculation and orientation. Score 0-30.
Role of Posttraumatic Stress Disorder at baseline on change in the percentage of heavy drinking days in preceding 4 weeks | Day 0
  Posttraumatic Stress Disorder Checklist for DSM-5 (PCL-5), a 17-item scale assessing the intensity of 17 PTSD symptoms. Each question is rated between 1 and 5 depending on the intensity and frequency of symptoms over the previous month. Three scales: Intrusion (items 1 to 5); Avoidance (items 6 to 12); Hyperstimulation (items 13 to 17). Total score 17-85, with threshold of 44 for PTSD diagnosis.
Role of attachment at baseline on change in the percentage of heavy drinking days in preceding 4 weeks | Day 0
  RSQ (Relationship Scale Questionnaire); a 30-item questionnaire classifying into four categories of attachment (secure or autonomous, avoidant or detached, preoccupied or ambivalent, fearful or disorganized). Score 13-65.
Change in the percentage of heavy drinking days in preceding 4 weeks according to concomitant Selective serotonin reuptake inhibitors | Day 0
  Concomitant Selective serotonin reuptake inhibitors yes/no
Change in the percentage of heavy drinking days in preceding 4 weeks according to concomitant Selective serotonin reuptake inhibitors | Week 3
  Concomitant Selective serotonin reuptake inhibitors yes/no
Change in the percentage of heavy drinking days in preceding 4 weeks according to concomitant Selective serotonin reuptake inhibitors | Week 6
  Concomitant Selective serotonin reuptake inhibitors yes/no
Change in the percentage of heavy drinking days in preceding 4 weeks according to concomitant Selective serotonin reuptake inhibitorsof other treatments on change in the percentage of heavy drinking days in preceding 4 weeks | Week 12
  Concomitant Selective serotonin reuptake inhibitors yes/no
Role of the patient-reported quality of the hallucinogenic experience on change in the percentage of heavy drinking days in preceding 4 weeks | End of 1st psilocybin session (Week 1)
  5D-ASC (5-Dimensional Altered States of Consciousness Questionnaire) dimension score after psilocybin sessions. A 94-item questionnaire (to be translated and retrotranslated) administered 5 to 6 hours after drug administration; visual analog scale of five main dimensions: "The absence of oceanic boundaries", "fear of ego dissolution", "restructuring of vision", "auditory alterations" and "reduction of vigilance".
Role of the patient-reported quality of the hallucinogenic experience on change in the percentage of heavy drinking days in preceding 4 weeks | End of 2nd psilocybin session (Week 4)
  5D-ASC (5-Dimensional Altered States of Consciousness Questionnaire) dimension score after psilocybin sessions. A 94-item questionnaire (to be translated and retrotranslated) administered 5 to 6 hours after drug administration; visual analog scale of five main dimensions: "The absence of oceanic boundaries", "fear of ego dissolution", "restructuring of vision", "auditory alterations" and "reduction of vigilance".
Role of the quality of the hallucinogenic experience according to brain activity on change in the percentage of heavy drinking days in preceding 4 weeks | Before 1st experimental session (Week 1)
  Electroencephalogram parameters: alpha coherence in the resting state
Role of the quality of the hallucinogenic experience according to brain activity on change in the percentage of heavy drinking days in preceding 4 weeks | During the 1st experimental session (Week 1)
  Electroencephalogram parameters: alpha coherence in the resting state
Role of the quality of the hallucinogenic experience according to brain activity on change in the percentage of heavy drinking days in preceding 4 weeks | Day after 2nd experimental session (Week 4)
  Electroencephalogram parameters: alpha coherence in the resting state
Change in the percentage of heavy drinking days in preceding 4 weeks according to the quality of the hallucinogenic experience | Day after 1st experimental session (Week 1)
  Hallucinogenic experience assessed through qualitative analysis of audio-recorded verbatim of the integration session.
Change in the percentage of heavy drinking days in preceding 4 weeks according to the quality of the hallucinogenic experience | Day after 2nd experimental session (Week 4)
  Hallucinogenic experience assessed through qualitative analysis of audio-recorded verbatim of the integration session.
immune profiles through the microbiota | day 0
  Evaluate participants' immune profiles in both groups through the microbiota before the first dose with circulating 16sDNA assay.
Evolution immune profiles through the microbiota | day 0
  Evaluate the evolution of the immune profiles of participants in both groups through the microbiota before the first dose with circulating 16sDNA assay.
Immune and inflammatory profiles using cerebral structural and functional MRI | day 0
  Evaluate the immune and inflammatory profiles in the 2 groups using cerebral structural and functional MRI prior to the first psilocybin administration.
Immune and inflammatory profiles using cerebral structural and functional MRI | week 3
  Evaluate the immune and inflammatory profiles in the 2 groups using cerebral structural and functional MRI 3 weeks after to the first psilocybin administration.
Evolution of Immune and inflammatory profiles using cerebral structural and functional MRI | day 0
  Evaluate the evolution of the immune and inflammatory profiles in the 2 groups using cerebral structural and functional MRI to the first psilocybin administration.
Evolution of Immune and inflammatory profiles using cerebral structural and functional MRI | week 3
  Evaluate the evolution of the immune and inflammatory profiles in the 2 groups using cerebral structural and functional MRI 3 weeks after to the first psilocybin administration.
immune profiles through the microbiota | week 3
  Evaluate participants' immune profiles in both groups through the microbiota before the first dose with circulating 16sDNA assay.
Evolution immune profiles through the microbiota | week 3
  Evaluate the evolution of the immune profiles of participants in both groups through the microbiota before the first dose with circulating 16sDNA assay.
Inflammatory profiles by measuring the cytokine TNF alpha in plasma | day 0
  Evaluate participants' inflammatory profiles in both groups through cytokine TNF alpha before the first dose. A tube of blood will be taken. The sample is transported to the laboratory at room temperature within 4 hours.
  Tubes are then centrifuged at 2000g for 10 min at room temperature, then aliquoted by 500µL into 1.5 mL Eppendorf LoBind Protein tubes for storage at -80°C prior to batch analysis.
Inflammatory profiles by measuring the cytokine TNF alpha in plasma | week 3
  Evaluate participants' inflammatory profiles in both groups through cytokine TNF alpha before the first dose. A tube of blood will be taken. The sample is transported to the laboratory at room temperature within 4 hours. Tubes are then centrifuged at 2000g for 10 min at room temperature, then aliquoted by 500µL into 1.5 mL Eppendorf LoBind Protein tubes for storage at -80°C prior to batch analysis.
analysis of intestinal microbiota : Number of species detected in the intestinal microbiota | day 0
  Patients will provide a stool sample, stored at -20°C and transported in an insulated bag to the hospital. The sample will be frozen at -80°C. The number of species detected in the intestinal microbiota will be recorded
analysis of intestinal microbiota : Number of species detected in the intestinal microbiota | week 3
  Patients will provide a stool sample, stored at -20°C and transported in an insulated bag to the hospital. The sample will be frozen at -80°C. The number of species detected in the intestinal microbiota will be recorded
analysis of intestinal microbiota : Distribution of species detected in the intestinal microbiota. | day 0
  Patients will provide a stool sample, stored at -20°C and transported in an insulated bag to the hospital. The sample will be frozen at -80°C. The distribution of the various bacterial species detected in the intestinal microbiota will be recorded
analysis of intestinal microbiota : Distribution of species detected in the intestinal microbiota. | week 3
  Patients will provide a stool sample, stored at -20°C and transported in an insulated bag to the hospital. The sample will be frozen at -80°C. The distribution of the various bacterial species detected in the intestinal microbiota will be recorded
analysis of intestinal microbiota : Diversity of species detected in the intestinal microbiota. | day 0
  Patients will provide a stool sample, stored at -20°C and transported in an insulated bag to the hospital. The sample will be frozen at -80°C. The diversity index according to the number of species will be recorded
analysis of intestinal microbiota : Diversity of species detected in the intestinal microbiota. | week 3
  Patients will provide a stool sample, stored at -20°C and transported in an insulated bag to the hospital. The sample will be frozen at -80°C. The diversity index according to the number of species will be recorded
Inflammatory profiles by measuring the cytokine IL-1b in plasma | day 0
  Evaluate participants' inflammatory profiles in both groups through cytokine IL-1b before the first dose. A tube of blood will be taken. The sample is transported to the laboratory at room temperature within 4 hours.
  Tubes are then centrifuged at 2000g for 10 min at room temperature, then aliquoted by 500µL into 1.5 mL Eppendorf LoBind Protein tubes for storage at -80°C prior to batch analysis.
Inflammatory profiles by measuring the cytokine IL-1b in plasma | week 3
  Evaluate participants' inflammatory profiles in both groups through cytokine IL-1b before the first dose. A tube of blood will be taken. The sample is transported to the laboratory at room temperature within 4 hours.
  Tubes are then centrifuged at 2000g for 10 min at room temperature, then aliquoted by 500µL into 1.5 mL Eppendorf LoBind Protein tubes for storage at -80°C prior to batch analysis.
Inflammatory profiles by measuring the cytokine IL-6 in plasma | day 0
  Evaluate participants' inflammatory profiles in both groups through cytokine IL-6 before the first dose. A tube of blood will be taken. The sample is transported to the laboratory at room temperature within 4 hours.
  Tubes are then centrifuged at 2000g for 10 min at room temperature, then aliquoted by 500µL into 1.5 mL Eppendorf LoBind Protein tubes for storage at -80°C prior to batch analysis.
Inflammatory profiles by measuring the cytokine IL-6 in plasma | week 3
  Evaluate participants' inflammatory profiles in both groups through cytokine IL-6 before the first dose. A tube of blood will be taken. The sample is transported to the laboratory at room temperature within 4 hours.
  Tubes are then centrifuged at 2000g for 10 min at room temperature, then aliquoted by 500µL into 1.5 mL Eppendorf LoBind Protein tubes for storage at -80°C prior to batch analysis.
Inflammatory profiles by measuring the cytokine IL-8 in plasma | day 0
  Evaluate participants' inflammatory profiles in both groups through cytokine IL-8 before the first dose. A tube of blood will be taken. The sample is transported to the laboratory at room temperature within 4 hours.
  Tubes are then centrifuged at 2000g for 10 min at room temperature, then aliquoted by 500µL into 1.5 mL Eppendorf LoBind Protein tubes for storage at -80°C prior to batch analysis.
Inflammatory profiles by measuring the cytokine IL-8 in plasma | week 3
  Evaluate participants' inflammatory profiles in both groups through cytokine IL-8 before the first dose. A tube of blood will be taken. The sample is transported to the laboratory at room temperature within 4 hours.
  Tubes are then centrifuged at 2000g for 10 min at room temperature, then aliquoted by 500µL into 1.5 mL Eppendorf LoBind Protein tubes for storage at -80°C prior to batch analysis.
Inflammatory profiles by measuring the cytokine IL-10 in plasma | day 0
  Evaluate participants' inflammatory profiles in both groups through cytokine IL-10 before the first dose. A tube of blood will be taken. The sample is transported to the laboratory at room temperature within 4 hours.
  Tubes are then centrifuged at 2000g for 10 min at room temperature, then aliquoted by 500µL into 1.5 mL Eppendorf LoBind Protein tubes for storage at -80°C prior to batch analysis.
Inflammatory profiles by measuring the cytokine IL-10 in plasma | week 3
  Evaluate participants' inflammatory profiles in both groups through cytokine IL-10 before the first dose. A tube of blood will be taken. The sample is transported to the laboratory at room temperature within 4 hours.
  Tubes are then centrifuged at 2000g for 10 min at room temperature, then aliquoted by 500µL into 1.5 mL Eppendorf LoBind Protein tubes for storage at -80°C prior to batch analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Amandine Luquiens, Principal Investigator — CHU de Nimes
Locations (1):
- CHU, Nîmes, Nîmes, France